CLINICAL TRIAL: NCT04645290
Title: Eficacia de Una intervención Multicomponente e Interdisciplinaria Sobre la Habilidad de Cuidado y Sobrecarga de Cuidadores Familiares de Personas Con Enfermedades crónicas Cardiocerebrovasculares
Brief Title: Efficacy of a Multicomponent and Interdisciplinary Intervention on the Care Ability and Burden of Family Caregivers of People With Chronic Cardiocerebrovascular Diseases
Acronym: Emiicare
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Claudia Aristizábal (Other)
Collaborators: Fundación Universitaria Sanitas (Unknown); Universidad Nacional de Colombia (Other); Universidad de Santander (Other)
Responsible Party: Sponsor-Investigator, Claudia Aristizábal, Coordinadora Unidad de Investigación, Sanitas University
Organization: Sanitas University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CEIFUS 389-19
Record Dates: First submitted 2020-11-05; First posted 2020-11-27 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Caregivers; Burnout, Psychological
Keywords: Cerebrovascular Disorders; Vascular Diseases; Treatment Outcome; Health Education; Interdisciplinary Research; Aptitud
MeSH Terms: conditions — Burnout, Psychological; Cerebrovascular Disorders; Vascular Diseases; Health Education

STUDY DESIGN:
Intervention Model Description: Double-blind controlled clinical trial-type experimental design , with a mixed approach (QUAN + qual), with an intervention group and a control group.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding of people in charge of both initial and final measurements, and of those who perform data analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: Educational Intervention "KARER" (Experimental): General objective of the intervention: Implement self-care strategies and care actions aimed at people facing chronic diseases with disabilities, applying knowledge, ability and attitudes that allow them to act in a timely manner, reducing the risk of complications, improving well-being and the quality of life of the person cared for and of himself. Through face-to-face, virtual interdisciplinary educational actions (B-learning) and with simulation support.
  Interventions: Behavioral: Intervention group: Educational Intervention "KARER"
- Usual Care (No Intervention): The people assigned to this group will receive their own responses from the institution providing care services to which they belong. These instructions consist of: information on the disease process and treatment received from the medical group, information on assistance by the nursing group and finally, the administrative procedures carried out by social work.

INTERVENTIONS:
Behavioral: Intervention group: Educational Intervention "KARER" — Multicomponent and interdisciplinary intervention on the care ability and burden of family caregivers. It consists of:
  Virtual componet
  * Module 0: the introduction
  * Module 1: called "Identifying my role as a caregiver"
  * Module 2: called "Strategies to strengthen care"
  * Module 3: called "Strengthening my caring skills"
  Face-to-face componed - Two seasons of 4 hours each
  Simulation component
  - One season of practices abilities of 4 hours.
  Other Names: Educational Intervention "Karer"
  Arms: Intervention group: Educational Intervention "KARER"

SUMMARY:
The purpose of this intervention is to improve the caregiving ability of family caregivers of people with cardiovascular diseases and therefore reduce burden caregiver through face-to-face, virtual interdisciplinary educational actions (B-learning) and with simulation support. The study will have two groups, one who will receive the intervention and the other with regular treatment.

DETAILED DESCRIPTION:
Introduction: In Colombia it is anticipated that demographic changes will have the effect of increasing the number of older adults who will require care by families, accompanied by a greater demand for institutional care services, due to the prevalence and confluence of various chronic non-communicable diseases (NCD) in this age group, where cardiocerebrovascular diseases especially stand out, which can additionally generate functional sequelae in the patient at a physical and cognitive level. The presence of specifically cardiocerebrovascular CNCD compromises the sick person and their family caregiver, who assumes this function within the home without receiving any type of economic remuneration, training, social support or any type of additional service offered by the system to cope with this role. Taking great importance the ability to care on the part of the caregivers of these people and its impact on their survival and on the management of the disease. Additionally, the events that frame the care of a person with NCD, added to the demand for direct care and the lack of social support, can trigger the family caregiver to present overload. Therefore, it is essential to create and implement interventions that promote the caregiving ability of family caregivers, from different approaches and perspectives, so that a multicomponent and interdisciplinary intervention becomes essential in this process.

Objective: To determine the efficacy of a multicomponent and interdisciplinary intervention in B-Learning modality and a clinical simulation component on the ability to care and the burden on family caregivers of people with chronic cardio-cerebral vascular diseases in a condition of disability, of home care programs and home hospitalization in the cities of Bogotá and Bucaramanga.

Method: a study with an experimental design type double-blind controlled clinical trial (blinding of the people in charge of both initial and final measurements, and of those who perform the data analysis), with a mixed approach (QUAN + qual), with a group intervention and a control group. The study will be carried out in the cities of Bogotá and Bucaramanga. For the collection of the information, the characterization format of sociodemographic and clinical variables will be used for family caregivers and people in their care, the Ngozi Nkongho care skill instrument and the Zarit care burden instrument, mainly. Similarly, participant observation will be carried out in face-to-face workshops where the body dimension is addressed as a means for the recognition of family caregivers, their abilities and achievements. Likewise, focus groups will be held at the end of each workshop with the caregivers who wish to participate, until the theoretical saturation is achieved. The analysis of quantitative data will include descriptive statistics, inferential analysis, and a repeated measures ANOVA to assess the intragroup and intergroup effects of the response variables. The analysis of the qualitative data will be carried out using content analysis techniques (coding) and grounded theory (open and axial coding), and then carry out a data triagulation within the method (qualitative), to complement the understanding of the phenomenon. study and as validation. Finally, a methodological triangulation (between methods) will be carried out based on the general objective of the study.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers aged 18 years or older.
* Be related to the person with cardiocerebrovascular disease in a condition of moderate to severe disability according to the Barthel scale.
* Having assumed the care of the person with a chronic illness in a condition of disability for a period greater than three months. (Note: if there is more than one family caregiver, the caregiver who has the longest stay in care and assistance will be selected).
* Know how to read and write.
* Have computer equipment and internet connectivity and a telephone
* Family caregivers residing in the cities of Bogotá and Bucaramanga.
* Accept voluntary participation in the study.

Exclusion Criteria:

* Family caregivers with cognitive and / or behavioral impairment that prevents them from participating in the research.
* Family caregivers of disabled people with cardiocerebrovascular disease, who are participating in other studies related to the topic of the research process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2022-03-20 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes of mean score ability from baseline at 2 months | baseline at 2 months
  It will measure with the "Caring Ability Inventory" (CAI): This instrument is composed of 37 items with a Likert-type graduation from 1 to 7, which are distributed in three subscales: knowledge, with 14 items, corage with 13 items, and patience with 10 items. The total score ranges from 37 to 259 points and the care ability is considered as: low (<203.1), medium (203.1 to 220.3), high (> 220.3).
Changes of mean score of burden caregivers from baseline at 2 months | baseline at 2 months
  It will measure with the "Zarit Burden Interview", The Zarit scale score ranges from 22 to 110 points and the caregiver burden is considered as: no burden (<or equal to 46), light burden (47 to 55), or heavy burden (> or equal to 56)

SECONDARY OUTCOMES:
Qualitative results: perception about caring ability and burden caregivers | one month
  Participant observation each face-to-face and simulation season and focal groups in the last face to face season: The participant observation will be carried out from the moment the face-to-face workshops begin, and will extend until the product of the observations is decreasing, that is, when the data begins to be repeated and no important new apprehensions are achieved.
  The focus groups will be held after the completion of the exploration and body expression workshops, with the participants who wish to do so. The context of the focus groups will be the same place of the workshop. It will be ensured that the focus groups do not last longer than 1 hour, in order not to interrupt the activities of family caregivers. The focus groups will be recorded in audio and will be transcribed as soon as they are held.
  This qualitative results will be focused in the perception of change experienced by the family caregivers about their caring ability and burden.

OTHER OUTCOMES:
Changes of the score of self-perceived health from baseline at 2 months | baseline at 2 months
  It will measure with the "The EQ-5D cuestionary": The EQ5D descriptive system is made up of five dimensions which are: 1) mobility, 2) self-care, 3) habitual activities, 4) pain or discomfort, and 5) anxiety and depression. These in turn are divided into five levels of perceived problems. A unique state of health is defined by combining one level from each of the five dimensions. In this way, a total of 3125 possible health states are defined. Each state is named by a 5-digit code. The second part of the instrument is made up of a visual analog scale from 0 to 100, the perception of the state of health at the time of measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Henry M Puerto Pedraza, RNs, MSc., Principal Investigator — Fundación Universitaria Sanitas
Locations (3):
- Colombia (3):
  - Fundación Universitaria Sanitas, Bogotá, Bogota D.C.
  - Universidad Nacional de Colombia, Bogotá, Bogota D.C.
  - Universidad de Santander, Bucaramanga, Santander Department

IPD SHARING:
Plan to Share IPD: No
Manuscript, Scientific Congress's, Share the results with the participants at the end of the research

REFERENCES:
- [Background] Nkongho, N. O. (2003). The caring ability inventory. Measurement of nursing outcomes, 3, 184-198
- [Background] Carrillo G GM, Sanchez-Herrera B, Barrera-Ortiz L. [Caring ability of family caregivers of children with cancer]. Rev Salud Publica (Bogota). 2015 May;17(3):394-403. doi: 10.15446/rsap.v17n3.32408. Spanish. PMID 28453089
- [Background] Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. Gerontologist. 1980 Dec;20(6):649-55. doi: 10.1093/geront/20.6.649. No abstract available. PMID 7203086
- See also: EQ-5D User Guides — https://euroqol.org/publications/user-guides/